CLINICAL TRIAL: NCT06001021
Title: The Effectiveness of Psychopharmacological Intervention Versus Cognitive Behavioral Couple Therapy and Their Combination in Perinatal Distressed Couples: A Randomized Clinical Trial
Brief Title: Cognitive Behavioral Couple Therapy for Perinatal Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameera Shafiq (Other)
Responsible Party: Sponsor-Investigator, Sameera Shafiq, Lecturer, University of Gujrat
Organization: University of Gujrat (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: UOG/ORIC/2022/393
Record Dates: First submitted 2023-06-26; First posted 2023-08-21 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Perinatal Depression; Perinatal Anxiety
Keywords: Cognitive Behavioral Couple Therapy (with or without Zikr); Pharmacology Intervention; Their combination

STUDY DESIGN:
Intervention Model Description: The first arm receives psychopharmacological medication. The second arm received CBCT (without Zikr). The third arm received CBCT (with Zikr). The fourth receives a combination of psychopharmacological medication and CBCT without Zikr The fifth arm receives a combination of psychopharmacological medication, CBCT, and with Zikr.
  The sixth control group receives either a placebo or no CBCT intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned to any of the above six arms by random number generation via online calculator.net. The outcome assessor (research assistant) will not be provided with information regarding the allocation of the participants to each group. Hence, the research assistant and participants will be blind to getting the questionnaires filled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Psychopharmacological Intervention (Experimental): This group will receive psychopharmacological intervention with perinatal safe light doses of antidepressants (see Langan et al., 2016; Schoretsanitis et al., 2021) and/or anxiolytic medications (see Nishimura et al, 2021; Saito et al, 2022) by a gynecologist. Selective Serotonin Reuptake Inhibitor (Escitalopram, 5-10 mg in pregnancy and Sertraline, 12.5-25 mg in postpartum) and/or Benzodiazepine (Alprazolam, 0.25-0.5 mg) will be prescribed in tablet form per day.
  Interventions: Drug: Psychopharmacological Intervention
- Cognitive Behavioral Couple Therapy (CBCT) Intervention (Experimental): This group will receive CBCT intervention from a trained psychologist in CBT. There are two conditions of CBCT, i) with Zikr, and ii) without Zikr.
  Interventions: Behavioral: Cognitive Behavioral Couple Therapy
- Combined Intervention (Experimental): This group will receive Medicine (prescribed by a consultant gynecologist) and CBCT intervention (with or without Zikr) from a trained psychologist in CBT.
  Interventions: Drug: Psychopharmacological Intervention; Behavioral: Cognitive Behavioral Couple Therapy; Other: Combination of Psychopharmacological Intervention and CBCT
- Control (Placebo and No Intervention) (Placebo Comparator): This group will receive a placebo from a gynecologist or no intervention from a trained psychologist.
  Interventions: Other: Placebo and No Intervention
- Other (No Intervention): This group will receive no intervention from a trained psychologist.

INTERVENTIONS:
Drug: Psychopharmacological Intervention — Escitalopram 5-10 mg in antenatal period; Sertraline 12.5-25 mg in postnatal period) and/or Benzodiazepine (Alprazolam, 0.25-0.50 mg).
  Arms: Combined Intervention; Psychopharmacological Intervention
Behavioral: Cognitive Behavioral Couple Therapy — CBCT intervention from a trained psychologist in CBT.
  Arms: Cognitive Behavioral Couple Therapy (CBCT) Intervention; Combined Intervention
Other: Combination of Psychopharmacological Intervention and CBCT — Medication will be prescribed by a consultant gynecologist and CBCT (conditions: with or without Zikr) will be provided by a trained psychologist.
  Arms: Combined Intervention
Other: Placebo and No Intervention — Control waitlist group will be provided with either a placebo by a consultant gynaecologist or no intervention by a trained psychologist
  Arms: Control (Placebo and No Intervention)

SUMMARY:
The hypotheses of the study are

* There will be differences in perceived perinatal distress, dyadic coping strategies, social support, domains of quality of life, and well-being in couples at Pre- and Post-Test levels during the perinatal period in couples.
* There will be differences with psychopharmacological intervention on total scores of perceived perinatal distress, dyadic coping strategies, social support, domains of quality of life, and well-being between the experimental and wait list-placebo control groups.
* There will be differences in CBCT (condition: without Zikr) on total scores of perceived perinatal distress, dyadic coping strategies, social support, domains of quality of life, and well-being between the experimental and wait list control group.
* There will be differences in CBCT (condition: with Zikr) on total scores of perceived perinatal distress, dyadic coping strategies, social support, domains of quality of life, and well-being between the experimental and wait list-placebo control groups.
* There will be differences for combined psychopharmacology, and CBT (conditions: with Zikr, without Zikr ) dimensions on total scores of perceived perinatal distress, dyadic coping strategies, social support, domains of quality of life, and well-being between experimental and wait list-placebo control group.

DETAILED DESCRIPTION:
The research questions of the study are

• How effective will psychopharmacological treatment, CBCT (with or without Zikr) and combined medicine-CBCT (with or without Zikr) interventions be in reducing symptoms of distress among couples during the perinatal period through a randomized clinical trial?

* Will dyadic coping strategies, social support, domains of quality of life, and well-being be improved in couples at the post-test level compared to the pre-test level by therapeutic intervention through a randomized clinical trial?
* What will be the effect size of post-test intervention?

Procedures and Protocol

The investigator will ask willing participants (screened for high risk) to select one of their preferred treatment modes out of the following

1. Medications (antidepressants and/or anxiolytics).
2. Cognitive Behavioural Therapy without Zikr.
3. Cognitive Behavioural Therapy with Zikr.
4. Combination of medications and cognitive behavioral therapy.
5. Combination of medications, cognitive behavioral therapy, and Zikr.

   A list of willing participants will be prepared. Each participant will have one in five chances of getting the preferred treatment mode after study is over. There will be two groups (experimental and control). To put people into one of the two groups, the investigator will select by randomization via online calculator random number generation.

   Participants will not know to which group they actually belong. This information will be recorded in the investigator's files, but the research assistant will not look at these files until after the research is finished. This is the best way the investigators have to testing without being influenced by what they think or hope might happen. Thus, the participants and the research assistant will be double blinded in the trial. The investigator and research assistant will then compare which of the two has the best results.

   The healthcare professionals (consultant gynecologists and investigator's research assistant) will be looking after the participants very carefully during the study. If there are anything participants are concerned about or that is bothering them about the research they will talk to the researcher, research assistant, gynaecologist or staff.

   A placebo or inactive medicine looks like real medicine but it is not. It is a dummy or pretend medicine. It has no effect on a person because it has no real medicine in it. The investigator wants to know whether medicine is good, therefore some people will be given the medicine and others will be given the pretend or a dummy medicine. For the research to be good, it is important that participants do not know whether they have been given real medicine or pretend or dummy medicine. This is one of the best ways the investigator have for knowing what the medicine that are being tested really does. But the participants given a placebo or no intervention will be informed at the end of the study and will be given treatment with medication as they are wait-list control. Moreover, the participants in the intervention group will receive their preferred treatment after the completion of the study.

   Participants will receive psychopharmacological treatment according to the National Institute for Health and Care Excellence (NICE) guidelines.

   Description of the Process

   During the research, a couple has to make ten visits to attend ten sessions in the hospital.

   • In the first visit, rapport will be built and pre-test assessment will be done in the following two approaches

   Quantitative Approach

   • Indigenously developed Parental Perinatal Distress Scale (PPDS).
   * Multidimensional Scale for Perceived Social Support (MSPSS).
   * Dyadic Coping Inventory (DCI).
   * Flourishing Scale (FS).
   * World Health Organization's Quality of Life Brief (WOLQOL-BREF)

   Qualitative Approach • In a qualitative approach, the semi-structured interviews will be conducted to explore the present stressors and expectations, and perceptions about the effectivity of treatments for perinatal distress among couples.

   Group 1 will be given medications or placebo for two weeks and/or for four to five weeks maximum (as per requirement) by the consultant gynaecologist. They have to visit after two weeks for post-test assessment. After treatment, the medicine will be tapered off to stop the intake. As explained before, neither participant will know whether they have received the medicine or the placebo. But in the end placebo participants will be debriefed and will be continued with real medication.

   Group 2, Group 3, Group 4 and Group 5 will continue the following 10 sessions (two sessions, each one hour per week) of CBCT with the investigator.

   • In the second session, participants will be psycho-educated for perinatal period distress, couples' physical and mental health and impact on the fetus-infant, the prevalence of depression and anxiety, and the significance of identification. Progressive muscle relaxation exercises will be carried out along with deep breathing. Feedback on the session will be taken.

   • In the third session, participants will be psycho-educated on the theoretical model of cognitive-behavioral couple therapy with some historical highlights and empirical standing. A thought log will be given for homework. Feedback for deep breathing and progressive muscle relaxation will be carried out.

   • In the fourth, fifth, sixth, seventh, eighth, and ninth session, feedback will be taken on homework and session. Various techniques of Cognitive Behavioural Couple Therapy will be applied based on the nature and contents of identified precipitating, perpetuating, and present stressors. In addition, relevant techniques will be incorporated from other modalities with eclecticism. Tasbeeh in Zikr will be given to group 3 and group 5 who opted for it in the screening process.

   • On the tenth visit, feedback on the session and homework will be taken. post-test assessment will be done in the following two approaches Group 6 will be exposed to one of the two conditions. 50% of couples will get a placebo and 50% will receive routine treatment care with no intervention. However, after the completion of the research, intervention groups and waitlist group (control) will be briefed and will be delivered with an intervention mode of treatment of their choice as selected earlier.

   Posttest assessment will be carried out by the following instruments Quantitative Approach • Indigenously developed Parental Perinatal Distress Scale (PPDS). • Multidimensional Scale for Perceived Social Support (MSPSS). • Dyadic Coping Inventory (DCI).

   • Flourishing Scale (FS).
   * World Health Organization's Quality of Life Brief (WOLQOL-BREF) Qualitative Approach
   * In a qualitative approach, the semi-structured interview will be conducted to explore the conception about the perinatal distress and perceptions about effectivity of treatments for perinatal distress among couples.

   Duration The research takes place from 15th August, 2023 to 30th September, 2023. Screening (for Major Depressive Disorder, Generalized Anxiety Disorder) with PPDS will be carried out on the couples who visit the gynecological ward of the hospital in August. After screening and signed informed consent, it will be necessary for participants to come to the clinic/hospital for 10 days in total, for one hour session each day in end of August and whole month of September (two sessions per week, each for one hour).

   The investigator and the research assistant would like to meet with participants twice in the upcoming month after the participant's last session visit for a final check-up in follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* The fourth month of pregnancy till the seventh month of the antenatal period.
* One week after delivery/birth till one year of a child in the postnatal period.
* Screened by PPDS as high-risk couples (for the level of severe symptomology) for Major Depressive Disorder (cut-off score 29 to 42) and/or Generalized Anxiety Disorder (cut-off score 17 to 24), and their Comorbidity.
* Dose requirements in any one of the antidepressant and/or anxiolytic, such as escitalopram (5-10 mg), sertraline (12.5-25 mg), and/or alprazolam (0.25-0.50 mg) per day.
* Wives accompanied by their husbands.
* Willingness to participate as a couple in the study.
* No physical disorder is present and/or no medication use.
* No psychiatric disorder history or presence
* No psychotropic medication use (presence or history)
* No disability is present.

Exclusion Criteria:

* Unwilling couples to participate in the study.
* Wife and/or couple is in an emergency.
* Wife and/or couple has unstable mental health.
* Wife accompanied by close relatives other than a spouse.
* Wife in the first week of delivery.
* Dose requirements in any one of the antidepressant and/or anxiolytic, such as escitalopram (above10 mg), sertraline (above 25 mg), and/or alprazolam (above 0.50 mg) per day.
* Couples screened with depressive disorder and/or anxiety disorder having psychotic features.
* Couples screened with depressive disorder and/or anxiety disorder having suicidal ideation.
* Couples screened with depressive disorder and/or anxiety disorder having mania/hypomanic features.
* Couples having diabetes.
* Couples having cardiovascular disorders.
* Presence or history of any physical or psychiatric disorder and/or use of medications
* Any intellectual, visual, or hearing disability present in either spouse of a couple.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Couples (wives and husbands)
Enrollment: 96 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gujrat, Gujrat, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langan R, Goodbred AJ. Identification and Management of Peripartum Depression. Am Fam Physician. 2016 May 15;93(10):852-8. PMID 27175720
- [Background] Schoretsanitis G, Westin AA, Stingl JC, Deligiannidis KM, Paulzen M, Spigset O. Antidepressant transfer into amniotic fluid, umbilical cord blood & breast milk: A systematic review & combined analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Apr 20;107:110228. doi: 10.1016/j.pnpbp.2020.110228. Epub 2021 Jan 2. PMID 33358964
- [Background] Nishimura A, Furugen A, Umazume T, Kitamura S, Soma M, Noshiro K, Takekuma Y, Sugawara M, Iseki K, Kobayashi M. Benzodiazepine Concentrations in the Breast Milk and Plasma of Nursing Mothers: Estimation of Relative Infant Dose. Breastfeed Med. 2021 May;16(5):424-431. doi: 10.1089/bfm.2020.0259. Epub 2021 Jan 15. PMID 33449825
- [Background] Saito J, Tachibana Y, Wada YS, Yakuwa N, Kawasaki H, Suzuki T, Sago H, Yamatani A, Murashima A. Transfer of brotizolam, periciazine, and sulpiride in cord blood and breast milk, and alprazolam in breast milk: a case report. J Pharm Health Care Sci. 2022 Apr 1;8(1):10. doi: 10.1186/s40780-022-00241-2. PMID 35361275
- [Background] Solmi M, Fornaro M, Ostinelli EG, Zangani C, Croatto G, Monaco F, Krinitski D, Fusar-Poli P, Correll CU. Safety of 80 antidepressants, antipsychotics, anti-attention-deficit/hyperactivity medications and mood stabilizers in children and adolescents with psychiatric disorders: a large scale systematic meta-review of 78 adverse effects. World Psychiatry. 2020 Jun;19(2):214-232. doi: 10.1002/wps.20765. PMID 32394557
- [Background] Yazdy MM, Mitchell AA, Louik C, Werler MM. Use of selective serotonin-reuptake inhibitors during pregnancy and the risk of clubfoot. Epidemiology. 2014 Nov;25(6):859-65. doi: 10.1097/EDE.0000000000000157. PMID 25171134
- [Background] Wilbraham D, Berg PH, Tsai M, Liffick E, Loo LS, Doty EG, Sellers E. Abuse Potential of Lasmiditan: A Phase 1 Randomized, Placebo- and Alprazolam-Controlled Crossover Study. J Clin Pharmacol. 2020 Apr;60(4):495-504. doi: 10.1002/jcph.1543. Epub 2019 Nov 20. PMID 31745991
- [Background] Pinheiro E, Bogen DL, Hoxha D, Ciolino JD, Wisner KL. Sertraline and breastfeeding: review and meta-analysis. Arch Womens Ment Health. 2015 Apr;18(2):139-146. doi: 10.1007/s00737-015-0499-y. Epub 2015 Jan 15. PMID 25589155
- [Background] Lee H, Koh JW, Kim YA, Chun KC, Han JY, Hwang JH, Choi JS, Joo SH, Kwon HY. Pregnancy and Neonatal Outcomes After Exposure to Alprazolam in Pregnancy. Front Pharmacol. 2022 Apr 25;13:854562. doi: 10.3389/fphar.2022.854562. eCollection 2022. PMID 35548333
- [Background] Petric D, Peitl MV, Peitl V. High doses alprazolam induced amenorrhoea and galactorrhoea. Psychiatr Danub. 2011 Mar;23(1):123-4. PMID 21448116
- [Background] Akhtar A, Rahman A, Husain M, Chaudhry IB, Duddu V, Husain N. Multidimensional scale of perceived social support: psychometric properties in a South Asian population. J Obstet Gynaecol Res. 2010 Aug;36(4):845-51. doi: 10.1111/j.1447-0756.2010.01204.x. PMID 20666955
- [Background] Bodenmann G. Dyadic coping inventory: Test manual. Bern, Switzerland: Huber. 2008.
- [Background] Choudhry FR, Al-Worafi YM, Akram B, Ahmed MA, Anwar Ul Haq M, Khan TM, Rehman IU, Barki N, Munawar K, Kamal A, Kassab YW, Bakrin FS, Golden KJ. Factor Structure of Urdu Version of the Flourishing Scale. Front Psychol. 2018 Sep 19;9:1513. doi: 10.3389/fpsyg.2018.01513. eCollection 2018. PMID 30283370
- [Background] Diener E, Wirtz D, Biswas-Diener R, Tov W, Kim-Prieto C, Choi DW, Oishi S. New measures of well-being. Assessing well-being: The collected works of Ed Diener. 2009:247-66.
- [Background] Saqib Lodhi F, Raza O, Montazeri A, Nedjat S, Yaseri M, Holakouie-Naieni K. Psychometric properties of the Urdu version of the World Health Organization's quality of life questionnaire (WHOQOL-BREF). Med J Islam Repub Iran. 2017 Dec 25;31:129. doi: 10.14196/mjiri.31.129. eCollection 2017. PMID 29951429
- [Background] Shafiq S, Bano Z, Randhawa SS, Khan KH, Muhammad QU, Muhammad A. Effectiveness of adapted cognitive behaviour therapy for dysthymia: An evidence based case study. J Pak Med Assoc. 2022 Mar;72(3):554-556. doi: 10.47391/JPMA.1412. PMID 35320244
- [Background] Shujja S, Adil A, Randall AK, Bodenmann G, Malik F. Psychometric properties and validity of Dyadic Coping Inventory-Urdu Version for use in Pakistan. Interpersona: An International Journal on Personal Relationships. 2020 Dec 22;14(2):183-99.
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Almurjan A, Macfarlane H, Badhan RKS. The application of precision dosing in the use of sertraline throughout pregnancy for poor and ultrarapid metabolizer CYP 2C19 subjects: A virtual clinical trial pharmacokinetics study. Biopharm Drug Dispos. 2021 Jun;42(6):252-262. doi: 10.1002/bdd.2278. Epub 2021 May 5. PMID 33851424
- [Background] Heinonen E, Blennow M, Blomdahl-Wetterholm M, Hovstadius M, Nasiell J, Pohanka A, Gustafsson LL, Wide K. Sertraline concentrations in pregnant women are steady and the drug transfer to their infants is low. Eur J Clin Pharmacol. 2021 Sep;77(9):1323-1331. doi: 10.1007/s00228-021-03122-z. Epub 2021 Mar 22. PMID 33751155
- [Background] Eichentopf L, Hiemke C, Conca A, Engelmann J, Gerlach M, Havemann-Reinecke U, Hefner G, Florio V, Kuzin M, Lieb K, Reis M, Riemer TG, Serretti A, Schoretsanitis G, Zernig G, Grunder G, Hart XM. Systematic review and meta-analysis on the therapeutic reference range for escitalopram: Blood concentrations, clinical effects and serotonin transporter occupancy. Front Psychiatry. 2022 Oct 17;13:972141. doi: 10.3389/fpsyt.2022.972141. eCollection 2022. PMID 36325531
- [Background] Bellantuono C, Bozzi F, Orsolini L. Safety of escitalopram in pregnancy: a case series. Neuropsychiatr Dis Treat. 2013;9:1333-7. doi: 10.2147/NDT.S45951. Epub 2013 Sep 9. PMID 24043940
- [Background] Bellantuono C, Bozzi F, Orsolini L, Catena-Dell'Osso M. The safety of escitalopram during pregnancy and breastfeeding: a comprehensive review. Hum Psychopharmacol. 2012 Nov;27(6):534-9. doi: 10.1002/hup.2265. Epub 2012 Oct 9. PMID 23044635

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychopharmacological Intervention: Escitalopram (5 mg) was prescribed by a gynecologist to high risk wives in antenatal period and to husbands in perinatal period.
  Sertraline (12.5 mg) was prescribed by a gynecologist to wives in the postnatal period.
- CBCT Intervention: 10 sessions each of 0ne hour, twice a week were carried out in group with the couples
- CBCT Intervention With Zikr: 10 sessions each of 0ne hour, twice a week were carried out in group with couples. Zikr (Ya Salam-The Peace Giver, Ya Rehman-The Merciful) was given for recitation.
- Combined Intervention Without Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk wives in the antenatal period and to husbands in the perinatal period. Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period. 10 sessions each of 0ne hour, twice a week were carried out in group with couples.
- Combined Intervention With Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk wives in the antenatal period and to husbands in the perinatal period. Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period. 10 sessions each of 0ne hour, twice a week were carried out in group with couples. Zikr (Ya Salam-The Peace Giver, Ya Rehman-The Merciful) were given for recitation.
- Control Arm (Placebo): In Placebo, sugar Pill was prescribed by a gynecologist.
- Control Arm (No Intervention): In no intervention, routine medical/gynecological checkups were carried out.
Period: 15 August 2023 to 30 September 2023
Arm/Group | Psychopharmacological Intervention | CBCT Intervention | CBCT Intervention With Zikr | Combined Intervention Without Zikr | Combined Intervention With Zikr | Control Arm (Placebo) | Control Arm (No Intervention)
Started | 16 | 16 | 16 | 16 | 16 | 8 | 8
Completed (These participants have completed the intervention and placebo/no intervention for the five primary outcomes of the study.) | 14 | 16 | 16 | 8 | 10 | 6 | 8
Not Completed | 2 | 0 | 0 | 8 | 6 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 8 | 6 | 2 | 0
Period: 1 October 2023 to 28 October 2023
Arm/Group | Psychopharmacological Intervention | CBCT Intervention | CBCT Intervention With Zikr | Combined Intervention Without Zikr | Combined Intervention With Zikr | Control Arm (Placebo) | Control Arm (No Intervention)
Started (Assessment of adverse events in the participants for the measurement of first secondary outcome) | 14 | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 8 | 10 | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable)
Completed (These participants have been assessed for the first secondary outcome (occurrence of adverse events) of the study.) | 14 | 0 | 0 | 8 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 1 October 2023 to 28 October 2023)
Arm/Group | Psychopharmacological Intervention | CBCT Intervention | CBCT Intervention With Zikr | Combined Intervention Without Zikr | Combined Intervention With Zikr | Control Arm (Placebo) | Control Arm (No Intervention)
Started (These participants have been assessed for the second secondary outcomes (blood concentration levels of escitalopram and sertraline) of the study.) | 14 | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 8 | 10 | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable) | 0 (Assessment of adverse events and blood concentration levels for escitalopram and sertraline in the participants is not applicable)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 0 | 0 | 8 | 10 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 0 | 0 | 8 | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Psychopharmacological Intervention: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
  Alprazolam (0.25 mg) is prescribed by a gynecologist to couples in antenatal and postnatal period.
- CBCT Without Zikr Intervention: 10 sessions each of 0ne hour, twice a week were carried out.
- CBCT With Zikr Intervention: 10 sessions each of 0ne hour, twice a week were carried out.
  Zikr (Ya Salam-The Peace Giver, Ya Rehman-The Merciful) was given for recitation.
- Combined Intervention Without Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
  Alprazolam (0.25 mg) is prescribed by a gynecologist to couples in antenatal and postnatal period.
  10 sessions each of 0ne hour, twice a week were carried out.
- Combined Intervention With Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
  Alprazolam (0.25 mg) is prescribed by a gynecologist to couples in antenatal and postnatal period.
  10 sessions each of 0ne hour, twice a week were carried out.
  Zikr (Ya Salam-The Peace Giver, Ya Rehman-The Merciful) were given for recitation.
- Placebo Comparator: Sugar Pill was prescribed by a gynecologist.
- No Intervention: Routine medical/gynecological checkups were carried out.
- Total: Total of all reporting groups
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention | Total
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.35 (3.83) | 30.37 (4.06) | 30.68 (4.98) | 30.50 (4.37) | 28.25 (3.01) | 34.33 (6.15) | 30.62 (2.97) | 30.56 (4.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 4 | 5 | 3 | 4 | 39
  Male | 7 | 8 | 8 | 4 | 5 | 3 | 4 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants] — All participants recruited in the present study were Asian Muslims, represented by participant flow count. "0" specified the absence of recruitment of the participants in a specified race.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 14 | 16 | 16 | 8 | 10 | 6 | 8 | 78
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Pakistan | 14 | 16 | 16 | 8 | 10 | 6 | 8 | 78
Absolute Value of Scores for High Risk Perinatal Distress (Anxiety and Depression) [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder Subscale and Major Depressive Disorder Subscale comprised 8 and 14 items respectively in Parental Perinatal Distress Scale. The response categories range from 0 to 3 scale. The total number of items in both subscales is 22. The summed scores obtained on 22 items ranged from 0 (minimum) to 66 (maximum). The high total score indicates worse symptoms of perinatal distress in the couples. In the present study, data mean and standard deviation specify absolute value at a pre-test treatment and post-test assessment.
  units on a scale | 60.21 (2.96) | 59.06 (3.15) | 59.18 (2.85) | 58.75 (3.28) | 52.70 (5.27) | 51.66 (2.33) | 59.62 (3.88) | 57.93 (4.41)
Absolute Value of Scores for Dyadic Coping Strategies [Mean (Standard Deviation); unit: units on a scale] — Dyadic Coping Inventory comprised 37 items with 1 to 5 scoring categories. However, items 36 and 37 were not included in the scoring as these were evaluative items. Scores for the remaining 35 items range from 35 (minimum) to 175 (maximum). The high score indicates better-than-average levels of coping skills in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in a pre-test and post-test assessment.
  units on a scale | 40.07 (2.26) | 38.87 (2.65) | 40.25 (2.56) | 42.50 (1.60) | 39.70 (2.90) | 40.66 (1.63) | 40.12 (1.64) | 40.11 (2.47)
Absolute Value of Scores for Perceived Social Support [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Scale for Perceived Social Support comprised 12 items. There are 1 to 7 scoring categories. The total scores range from 12 (minimum) to 84 (maximum). The high score indicates better social support for perinatal couples. In the present study, data mean and standard deviation specifies absolute values in a pre-test and post-test assessment.
  units on a scale | 20.07 (3.02) | 20.06 (2.76) | 18.31 (1.99) | 21.00 (2.00) | 17.50 (1.58) | 19.16 (3.31) | 18.87 (2.03) | 19.28 (2.59)
Absolute Value of Scores for Wellbeing [Mean (Standard Deviation); unit: units on a scale] — The Flourishing Scale comprised 8 items with 1 to 7 scoring categories. Scores range from 8 (minimum) to 56 (maximum). The high score indicates better well-being in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in a pre-test and post-test assessment.
  units on a scale | 11.14 (2.07) | 11.12 (2.12) | 10.50 (2.28) | 11.37 (1.68) | 9.80 (1.75) | 10.33 (1.63) | 9.87 (1.64) | 10.66 (1.99)
Absolute Value of Scores for Physical Subscale of World Health Organization Quality of Life Bref [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Bref (WHOQOL-BREF) comprised 26 items with 1 to 5 scoring categories.
  Evaluative items 1 and 2 were not included in the scoring. The remaining 24 items are classified in four subscales (physical, psychological, social, environmental) of quality of life. Scores for physical subscale (7 items) ranged from 7 (minimum) to 35 (maximum). The high score indicates a better physical quality of life in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in a pre-test and post-test assessment.
  units on a scale | 9.21 (1.36) | 9.75 (1.23) | 9.56 (1.31) | 10.62 (0.91) | 9.70 (1.33) | 9.66 (0.81) | 9.37 (1.59) | 9.65 (1.28)
Absolute Value of Score for Psychological Subscale of World Health Organization Quality of Life Bref [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Bref (WHOQOL-BREF) comprised 26 items with 1 to 5 scoring categories.
  Evaluative items 1 and 2 were not included in the scoring. The remaining 24 items are classified in four subscales (physical, psychological, social, environmental) of quality of life. Scores are 6 (minimum) to 30 (maximum) for psychological subscale (6 items). The high score indicates a better quality of life in psychological domain of perinatal couples. In the present study, data mean and standard deviation specifies absolute values in pre-test and post-test assessment.
  units on a scale | 8.500 (1.09) | 7.93 (1.28) | 8.93 (0.92) | 9.25 (0.70) | 8.90 (0.99) | 9.16 (0.75) | 8.50 (0.92) | 8.65 (1.07)
Absolute Value of Scores for Social Subscale of World Health Organization Quality of Life Bref [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Bref (WHOQOL-BREF) comprised 26 items with 1 to 5 scoring categories.
  Evaluative items 1 and 2 were not included in the scoring. The remaining 24 items are classified in four subscales (physical, psychological, social, environmental) of quality of life. Scores 3 (minimum) to 20 (maximum) are for social subscale (3 items). The high score indicates a better social quality of life in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in pre-test and post-test assessment.
  units on a scale | 3.50 (0.61) | 3.87 (0.61) | 3.43 (0.62) | 3.75 (0.70) | 3.70 (0.48) | 3.50 (0.54) | 4.00 (0.75) | 3.66 (0.61)
Absolute Value of Scores for Environment Subscale of World Health Organization Quality of Life Bref [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Bref (WHOQOL-BREF) comprised 26 items with 1 to 5 scoring categories.
  Evaluative items1 and 2 were not included in the scoring. The remaining 24 items are classified in four subscale (physical, psychological, social, environmental) of quality of life. Scores ranged 8 (minimum) to 40 (maximum) for environmental subscale (8 items). The high score indicates a better environmental quality of life in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in pre-test and post-test assessment.
  units on a scale | 9.28 (1.06) | 8.68 (0.79) | 9.68 (0.79) | 10.25 (0.88) | 9.40 (0.96) | 10.00 (0.89) | 9.00 (1.19) | 9.38 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: The Sum of Scores of Major Depressive Disorder Subscale and Generalized Anxiety Disorder Subscale
Description: The Generalized Anxiety Disorder Subscale and Major Depressive Disorder Subscale comprised 8 and 14 items respectively in Parental Perinatal Distress Scale. The response categories range from 0 to 3 scale. The total number of items in both subscales is 22. The summed scores obtained on 22 items range from 0 (minimum) to 66 (maximum). The high total score indicates worse symptoms of perinatal distress in the couples. In the present study, data mean and standard deviation specify absolute value at a pre-test and post-test assessment.
Time Frame: After recruitment, screening, randomization, and allocation, Pre-test Assessment on week 1 (Baseline Measures) and post-test assessment on week 10 (Outcome Measures) through the study period completion.
Population: The target enrollment was met and planned statistical analyses were performed. The impact of treatment (psychopharmacological medicine; CBCT; CBCT along with Zikr; combined (Psychopharmacological medicine and CBCT); combined (Psychopharmacological and CBCT along with Zikr), placebo comparator, and no intervention is measured for perinatal distress via ANCOVA after controlling for baseline pre-test scores for perinatal distress (depression and anxiety) and monthly income in SPSS-24.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Psychopharmacological Intervention: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
- CBCT With Zikr Intervention: 10 sessions each of 0ne hour, twice a week were carried out. Zikr (Ya Salam-The Peace Giver, Ya Momin-The Faith Giver, Ya Rehman-The Merciful) was given for recitation.
- Combined Intervention Without Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
  10 sessions each of 0ne hour, twice a week were carried out.
- Combined Intervention With Zikr: Escitalopram (5 mg) is prescribed by a gynecologist to high-risk couples in the antenatal period and to husbands in the postnatal period.
  Sertraline (12.5 mg) is prescribed by a gynecologist to women in postnatal period.
  10 sessions each of 0ne hour, twice a week were carried out.
  Zikr (Ya Salam-The Peace Giver, Ya Rehman-The Merciful) were given for recitation.
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8
score on a scale | 18.14 (2.03) | 17.31 (2.33) | 15.62 (2.47) | 8.62 (1.50) | 9.50 (1.35) | 53.33 (2.87) | 60.12 (4.12)
Statistical Analysis 1: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Test type: Superiority — In the Superiority Trial, the statistical test aims to show that the treatment group gives better results than the control group. In an equivalence trial, the statistical test aims to show that two treatments are not too different in characteristics, where "not too different" is defined in a clinical manner (Lesaffre, 2008). Lesaffre E. Superiority, equivalence, and non-inferiority trials. Bull NYU Hosp Jt Dis. 2008;66(2):150-4. PMID: 18537788; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = -35.55, 90% CI 2-sided [-38.90 to -32.19], Standard Deviation 17.78

2. Primary Outcome: The Sum of Scores on Multidimensional Scale for Perceived Social Support (MSPSS)
Description: The Multidimensional Scale for Perceived Social Support comprised 12 items. There are 1 to 7 scoring categories. The sum of score for 12 items range from 12 (minimum) to 84 (maximum). The high score indicates better social support for perinatal couples. In the present study, data mean and standard deviation specifies absolute values in post-test assessment.
Time Frame: as for outcome 1
Population: The target enrollment was met and planned statistical analyses were performed. The impact of treatment (psychopharmacological medicine; CBCT; CBCT along with Zikr; combined (Psychopharmacological medicine and CBCT); combined (Psychopharmacological and CBCT along with Zikr), placebo comparator, and no intervention is measured for perceived social support via ANCOVA after controlling for baseline pre-test scores for perinatal distress (depression and anxiety) and monthly income in SPSS-24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8
score on a scale | 22.14 (1.40) | 38.31 (4.40) | 47.00 (2.00) | 79.00 (3.20) | 80.50 (2.63) | 18.66 (3.32) | 18.62 (1.59)
Statistical Analysis 1: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 23.96, 90% CI 2-sided [19.59 to 28.32], Standard Deviation 23.14

3. Primary Outcome: The Sum of Scores on Dyadic Coping Inventory (DCI)
Description: Dyadic Coping Inventory comprised 37 items with 1 to 5 scoring categories. However, items 36 and 37 were not included in the scoring as these were evaluative items. The sum of scores for the remaining 35 items range from 35 (minimum) to 175 (maximum). The high score indicates better-than-average levels of coping skills in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in post-test assessment.
Time Frame: as for outcome 1
Population: The target enrollment was met and planned statistical analyses were performed. The impact of treatment (psychopharmacological medicine; CBCT; CBCT along with Zikr; combined (Psychopharmacological medicine and CBCT); combined (Psychopharmacological and CBCT along with Zikr), placebo comparator, and no intervention is measured for dyadic coping via ANCOVA after controlling for baseline pre-test scores for perinatal distress (depression and anxiety) and monthly income in SPSS-24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8
score on a scale | 105.42 (2.97) | 153.25 (1.77) | 155.93 (3.83) | 161.37 (3.24) | 162.40 (4.90) | 41.16 (1.16) | 40.25 (1.48)
Statistical Analysis 1: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.00, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 86.89, 90% CI 2-sided [78.33 to 95.46], Standard Deviation 45.43

4. Primary Outcome: The Sum of Scores on Flourishing Scale (FS)
Description: The Flourishing Scale comprised 8 items with 1 to 7 scoring categories. Sum of scores range from 8 (minimum) to 56 (maximum) for eight items. The high score indicates better well-being in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in pre-test and post-test assessment.
Time Frame: as for outcome 1
Population: The target enrollment was met and planned statistical analyses were performed. The impact of treatment (psychopharmacological medicine; CBCT; CBCT along with Zikr; combined (Psychopharmacological medicine and CBCT); combined (Psychopharmacological and CBCT along with Zikr), placebo comparator, and no intervention is measured for perceived wellbeing via ANCOVA after controlling for baseline pre-test scores for perinatal distress (depression and anxiety) and monthly income in SPSS-24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8
score on a scale | 19.78 (3.40) | 38.56 (1.89) | 38.31 (2.33) | 52.37 (2.97) | 50.80 (2.57) | 9.83 (1.60) | 9.50 (1.51)
Statistical Analysis 1: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 22.26, 90% CI 2-sided [19.41 to 25.12], Standard Deviation 15.15

5. Primary Outcome: The Sum of Scores on Each Subscale of World Health Organization Quality of Life (WHOQOL-BREF)
Description: World Health Organization Quality of Life Bref (WHOQOL-BREF) comprised 26 items with 1 to 5 scoring categories. Item 1 and item 2 were not included in the scoring domains because these were evaluative items. The remaining 24 items are classified in four subscales (physical, psychological, social, and environmental) of quality of life. Sum of scores for physical aspect (7 items) of life ranged from 7 (minimum) to 35 (maximum); 6(minimum) to 30 (maximum) for psychological subscale (6 items); 3 (minimum) to 20 (maximum) for social subscale(3 items); and 8 (minimum) to 40 (maximum) for environmental subscale (8 items) of life. The high score indicates a better quality of life in that particular subscale domain in perinatal couples. In the present study, data mean and standard deviation specifies absolute values in pre-test and post-test assessment.
Time Frame: as for outcome 1
Population: Target enrollment was met, planned statistical analyses were performed. The impact of treatment (psychopharmacological; CBCT; CBCT along with Zikr; combined (Psychopharmacological and CBCT); combined (Psychopharmacological and CBCT along with Zikr), placebo comparator, and no intervention is measured for physical, psychological, social, and environmental quality of life via ANCOVA after controlling for pre-test scores for perinatal distress (depression and anxiety) and monthly income in SPSS-24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 16 | 16 | 8 | 10 | 6 | 8
score on a scale
  Post Test Assessment on Physical Subscale | 29.07 (2.12) | 29.12 (2.02) | 30.06 (3.02) | 29.50 (2.07) | 30.20 (1.93) | 10.00 (0.89) | 10.50 (1.41)
  Post Test Assessment on Psychological Subscale | 28.64 (1.08) | 28.37 (1.20) | 29.06 (0.92) | 28.75 (1.03) | 28.80 (1.22) | 9.66 (0.51) | 9.25 (0.70)
  Post Test Assessment on Social Subscale | 13.50 (0.75) | 13.56 (0.96) | 13.93 (0.92) | 13.50 (0.92) | 13.90 (0.99) | 3.66 (0.99) | 4.12 (0.64)
  Post Test Assessment on Environmental Subscale | 37.92 (1.14) | 38.31 (1.13) | 38.18 (1.10) | 37.87 (1.12) | 38.70 (0.94) | 10.16 (0.75) | 9.62 (0.74)
Statistical Analysis 1: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Physical Domain of Quality of Life; Test type: Superiority — In the Superiority Trial, the statistical test aims to show that the treatment group gives better results than the control group. In an equivalence trial, the statistical test aims to show that two treatments are not too different in characteristics, where "not too different" is defined in a clinical manner (Lesaffre, 2008); p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 16.44, 90% CI 2-sided [15.02 to 17.87], Standard Deviation 7.55
Statistical Analysis 2: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Psychological Domain of Quality of Life; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 16.60, 90% CI 2-sided [15.16 to 18.04], Standard Deviation 7.62
Statistical Analysis 3: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Social Domain of Quality of Life; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 8.26, 90% CI 2-sided [7.52 to 9.01], Standard Deviation 3.96
Statistical Analysis 4: Comparison: Psychopharmacological Intervention vs CBCT Without Zikr Intervention vs CBCT With Zikr Intervention vs Combined Intervention Without Zikr vs Combined Intervention With Zikr vs Placebo Comparator vs No Intervention; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.000, ANCOVA — The significance level is 0.10 with 90% confidence interval; Mean Difference (Final Values) = 23.73, 90% CI 2-sided [21.64 to 25.81], Standard Deviation 11.07

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Side effects of escitalopram and sertraline (5 mg/day, and 12.5 mg/day respectively) classified as Grade 1 level in CTCAE v4.0 as these settle down within two to three weeks of medication. A checklist assessed presence or absence of adverse events among participants in psychopharmacological intervention arm, combined intervention without zikr arm, and combined intervention with zikr arm qualitatively. The overall number of participants analyzed in Secondary Outcome Period Participants (1st Oct to 28 Oct) represent the total number of participants for whom an Outcome Measure was measured and analyzed from the Primary Outcome Period Participants, for each Arm/Group. The data were not collected and the outcome cannot be reported for arms without psychopharmacological intervention including "0" participants analyzed because medication was not administered.
Time Frame: After recruitment, screening, randomization, and allocation, number of participants with treatment-related adverse events as assessed by CTCAE v4.0 on week 11 and week 12 (follow-ups) through the study period (two and half months).
Population: Adverse events (AE) were not assessed for CBCT (Without or With Zikr), Placebo & No Intervention Arms; 0 specified absence. AE were assessed systematically with checklist in psychopharmacology & combined arms (with, without Zikr); Zero specified absence of all-cause mortality and serious AE. Total Number of Participants at Risk showed Participant Flow module count. Other (non-serious) AE, mild transitional side effects (nausea, stomachache) were reported with frequency threshold above 5%.
Measure: Count of Participants; unit: Participants
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 14 | 0 | 0 | 8 | 10 | 0 | 0
Participants
  Other [Not Including Serious] Adverse Events: Nausea | 2 | 0 | 0 | 1 | 1 | 0 | 0
  Other [Not Including Serious] Adverse Events: Stomach Pain | 1 | 0 | 0 | 1 | 1 | 0 | 0

7. Secondary Outcome: Changes in Blood Concentration (Either ng/ml or mg/L) Levels for Escitalopram and Sertraline
Description: Gynaecologist prescribed 5 mg/day escitalopram antenatally or 12.5 mg/day sertraline postnatally. Assessment of blood concentration level via High Performance Liquid Chromatography was conditioned on consent of the participants. The overall number of participants analyzed in Secondary Outcome Period Participants (1st Oct to 28 Oct) represent the total number of participants from the Primary Outcome Period, for each Arm/Group. The data were not collected and the outcome cannot be reported for arms without psychopharmacological intervention including "0" participants. The participants withdrew from HPLC to avoid expansive biomedical tests, adhering to Pakistani cultural norm. The toxicity levels is not reported in the blood of the couples because 5 mg/day escitalopram (Eichentopf et al; Bellantuono et al) or 12.5 mg/day sertraline (Almurjan et al ; Heinonen et al) and is considered safe dose range with no sign of toxicity in blood concentration levels and no presence of adverse events.
Time Frame: After recruitment, screening, randomization, and allocation, changes in blood concentration levels for Escitalopram and Sertraline as assessed on week 12 (follow-up) through the study period (two and half months).
Population: No medicine was prescribed in CBCT (with, without Zikr), placebo, and no intervention arms and "N/A" indicate absence of assessment in these arms. The subjects withdraw from blood test consent in psychopharmacological arm, combined intervention with zikr arm, and combined intervention without zikr arm and "Zero" specified the absence of assessment of blood concentration levels (5 mg escitalopram or 12.5 mg sertraline) due to participants' withdrawal.
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was assessed on week 11 and week 12 (follow-ups) through the study period (2 and half months).
Description: Definition of adverse events did not differ from the clinicaltrials.gov Definitions. Total Number of Participants at Risk for adverse events were not assessed for "CBCT Without Zikr", "CBCT With Zikr", "Placebo Comparator" and "No Intervention" Arms. "N/A" specified absence of assessment for the participants.
  In psychopharmacology, combined arms no all-cause mortality and serious adverse event was observed, represented by zero. Total Number of Participants at Risk showed Participant Flow count.
Arm/Group | Psychopharmacological Intervention | CBCT Without Zikr Intervention | CBCT With Zikr Intervention | Combined Intervention Without Zikr | Combined Intervention With Zikr | Placebo Comparator | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/0 | 0/0 | 0/8 | 0/10 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/0 | 0/0 | 0/8 | 0/10 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/14 | 0/0 | 0/0 | 2/8 | 2/10 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychopharmacological Intervention (N=14) | CBCT Without Zikr Intervention (N=0) | CBCT With Zikr Intervention (N=0) | Combined Intervention Without Zikr (N=8) | Combined Intervention With Zikr (N=10) | Placebo Comparator (N=0) | No Intervention (N=0)
Serious Adverse Event (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Serious Adverse Event (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serious Adverse Event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychopharmacological Intervention (N=14) | CBCT Without Zikr Intervention (N=0) | CBCT With Zikr Intervention (N=0) | Combined Intervention Without Zikr (N=8) | Combined Intervention With Zikr (N=10) | Placebo Comparator (N=0) | No Intervention (N=0)
Other (Not including Serious) Adverse Events (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not Including Serious) Adverse Event terms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not including Serious) Adverse Events (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not Including Serious) Adverse Event terms (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not Including Serious) Adverse Event terms (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (Not Including Serious) Adverse Event terms (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT06001021/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT06001021/SAP_001.pdf
  • Informed Consent Form (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT06001021/ICF_002.pdf